CLINICAL TRIAL: NCT01788696
Title: Assessment of the Effect of Treatment Pathways, Adherence, and Treatment Efficacy in Parkinson's Disease Subjects Randomized to SPECT Imaging of the Dopamine Transporter (Ioflupane I123 Injection)
Brief Title: Pilot Study To Assess Effect of Treatment and Adherence in PD Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00036503
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson Disease
Keywords: Parkinsonism; Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Early Imaging (Active Comparator): Group A will receive SPECT imaging 3 times during the study. The first scan will take place prior to the initiation of any treatment, followed by scans at week 26 and week 52.
  Interventions: Radiation: Group A - Early Imaging
- Group B - Delayed Imaging (Active Comparator): Group B will receive SPECT imaging 2 times during the study. Group B will not have the first scan (prior to the initiation of any treatment). Scan will take place at week 26 and week 52.
  Interventions: Radiation: Group B - Delayed Imaging

INTERVENTIONS:
Radiation: Group A - Early Imaging — Total of 3 scans
  Other Names: [123I]-FP-CIT SPECT
  Arms: Group A - Early Imaging
Radiation: Group B - Delayed Imaging — Total of 2 scans
  Other Names: [123I]-FP-CIT SPECT
  Arms: Group B - Delayed Imaging

SUMMARY:
The purpose of this study is to evaluate the impact of imaging the brain as a diagnostic tool in the management of early Parkinson's disease (PD).

DETAILED DESCRIPTION:
The imaging drug used in this study is Ioflupane (123I) Injection, also referred to as DaTscan. DaTscan is FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80;
* diagnosis of idiopathic PD exhibiting at least 2 of 3 cardinal signs (bradykinesia, rigidity and resting tremor);
* maximum duration of previous exposure to anti-parkinsonian therapy being < 8 weeks;
* ability to signed informed consent;
* willingness and ability to complete medication diary and questionnaires;
* if a female subject of child-bearing potential, the use of an effective method of contraception.

Exclusion Criteria:

* current treatment with anti-parkinsonian medication;
* previous treatment with anti-parkinsonian medication for greater than 8 weeks;
* inability to complete questionnaires;
* unwillingness to complete all questionnaires and medication diary;
* subjects with secondary causes of parkinsonism;
* participant has evidence of clinical significant thyroid disease, gastrointestinal, cardiovascular, hepatic, renal, hematologic, neoplastic, endocrine, neurologic, immunodeficiency, pulmonary, or other medical or psychiatric disorder;
* positive serum/urine pregnancy test at any time during the study period;
* the participant has a history of alcohol, narcotic, or any other drug abuse as defined by the DSM-IV within the past 2 years;
* participation in a concurrent PD trial within 60 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Patient adherence to treatment plan | 1 year
  Patient and treating physician agree on a treatment plan at visit 3. Patient adherence to medications will be evaluated based on pill count at each follow-up study visit. Additionally, each patient will record their adherence to therapy on the Patient Expectations and Disease-related Questionnaire (PEDQ) at each follow-up study visit, allowing the study team to track compliance with pharmacologic therapy as well as treatments including therapy exercise plans.

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS) | 1 year
  Other outcome measures will be between any group differences in UPDRS.
Life Orientation Test - Revised (LOT-R) | 1 year
  Other outcome measures will be between any group differences in LOT-R. This test assesses individual differences in generalized optimism versus pessimism.
Marlowe - Crowne Social Desirability Scale (MCSD) | 1 year
  Other outcome measures will be between any group differences in MCSD. This test assesses the extent to which individuals attempt to depict themselves as similar to the norms and standards of their society and community.
Obsessive - Compulsive Inventory (OCI) | 1 year
  Other outcome measures will be between any group differences in OCI. This self-report scale assesses distress from symptoms commonly experienced in obsessive-compulsive disorder.
Expectation of Global Response (EGCR) | 1 year
  Other outcome measures will be between any group differences in EGCR.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hickey, DO, Principal Investigator — Duke University Health Center
Locations (1):
- Duke University Health Center, Durham, North Carolina, United States